CLINICAL TRIAL: NCT05308342
Title: Clinical Study of Human Umbilical Cord Mesenchymal Stem Cells in the Treatment of Premature Ovarian Insufficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Li-jun Ding (Other)
Responsible Party: Sponsor-Investigator, Li-jun Ding, principal investigator, Nanjing University
Organization: Nanjing University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SZ-POF-2019-4
Record Dates: First submitted 2019-11-25; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Premature Ovarian Insufficiency
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UC-MSCs+hormone replacement group (Experimental): Group A was the hormone replacement combined with transplantation of umbilical cord mesenchymal stem cells group(test group).
  Interventions: Procedure: transplantation of human UC-MSCs into ovaries of POI patients; Drug: hormone replacement treatment
- hormone replacement group (Active Comparator): Group B was the hormone replacement group (control group).
  Interventions: Drug: hormone replacement treatment

INTERVENTIONS:
Procedure: transplantation of human UC-MSCs into ovaries of POI patients — UC-MSCs (GMP grade, from Clinical Center for Stem Cell Research of the Affiliated Drum Tower Hospital of Nanjing University Medical School, licensed by the China Food and Drug Administration) are injected into the ovary of patients under transvaginal ultrasonographic (TVUS)-guidance. A total number of 10×106 cells, 5×106 for unilateral ovarian injection) is immediately preserved and transferred for direct injection. After vaginal sterilization, TVUS-guided transplantation is performed by two senior-level medical physicians, using a SIEMENS ACUSON ANTANES premium edition system (SIEMENS AG Healthcare Sector, Erlangen, Germany), equipped with a 6-10 MHz probe. The UC-MSC solution is injected into the ovary by using 21-G PTC needles (Hakko Medical Co, Japan) under TVUS guidance.
  Arms: UC-MSCs+hormone replacement group
Drug: hormone replacement treatment — Routine estrogen progesterone replacement periodic therapy
  Other Names: HRT

SUMMARY:
This study was a single-center, randomized, controlled prospective study. Those who had premature ovarian failure and who had fertility requirements were enrolled in the study. To determine the efficacy and safety of umbilical cord mesenchymal stem cells in the treatment of patients with POI.

DETAILED DESCRIPTION:
According to the enrollment and exclusion criteria, the patients were enrolled, and the subjects were randomly divided into two groups by computer randomization. Group A was hormone replacement combined with transplantation of umbilical cord mesenchymal stem cells (test group). Group B was the hormone replacement group (control group).

ELIGIBILITY:
Inclusion Criteria:

1. Those who meet the POF diagnostic criteria and have no spontaneous follicular activity;
2. Married, 20 years old ≤ age < 40 years old;
3. The average diameter of each ovary is > 10 mm;
4. Have agreed to sign the informed consent form.

Exclusion Criteria:

1. Female and/or male chromosomal abnormalities;
2. Endometriosis, adenomyosis;
3. Postoperative ovarian borderline or malignant tumor;
4. Uterine dysplasia;
5. Associated with female autoimmune disease or other serious internal surgical diseases;
6. hormone replacement contraindications;
7. In the past 1 year, had received an experimental study of premature ovarian failure in the external hospital;
8. Male azoospermia or severe oligozoospermia.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Follicular development rate | 9-12 months
  Follicular development and hormonal examination were performed 1 week before treatment and at 1, 2, and 3 weeks after treatment to evaluate the development of follicles. If there is no follicular development in the third week, stop the drug after 1 week, and contact the next treatment time after menstruation. During the follow-up period to half a year after the end of the last treatment, the follicular development activity rate was observed.

SECONDARY OUTCOMES:
Changes in blood flow index in the ovary | 9-12 months
  Ovarian artery blood flow spectrum PI; RI; S/D (L; R)
Clinical pregnancy rate | 9-12 months
  Clinical pregnancy was defined as diagnosed by increasing serum concentration of beta-HCG 14 days after embryo transfer, and the subsequent demonstration of an intrauterine gestational sac by ultrasonography on 30 days after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Guangshu Han, phD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Reproductive Medicine Center, The affiliated Drum Towel Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China